CLINICAL TRIAL: NCT05415423
Title: Developing an Objective Measure of Experienced Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-00236
Record Dates: First submitted 2022-05-30; First posted 2022-06-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pain, Acute
Keywords: Measurement of Pain; Pain
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Study 1 Low-Intensity Group (Active Comparator): Control group which receives less intense electrical stimuli than the other.
  Interventions: Behavioral: Developing an objective measure of experienced pain
- Study 1 High-Intensity Group (Experimental): Group which receives more intense electrical stimuli than the other.
  Interventions: Behavioral: Developing an objective measure of experienced pain
- Study 2 Low-Intensity Group (Active Comparator): Control group which receives less intense heat stimuli than the other.
  Interventions: Behavioral: Developing an objective measure of experienced pain
- Study 2 High-Intensity Group (Experimental): Group which receives more intense heat stimuli than the other.
  Interventions: Behavioral: Developing an objective measure of experienced pain
- Study 3 Placebo group (Placebo Comparator): A group that receives a placebo cream.
  Interventions: Behavioral: Developing an objective measure of experienced pain
- Study 3 Painkiller group (Experimental): A group that receives a topical analgesic such as EMLA cream.
  Interventions: Behavioral: Developing an objective measure of experienced pain
- Study 4 test-retest reliability group (No Intervention): Participants who participated in either Study 1 or 2 are recruited. They will experience both electrical and heat stimuli.

INTERVENTIONS:
Behavioral: Developing an objective measure of experienced pain — At the beginning of each study, participants are randomly allocated into one of two groups.
  Within each group all participants are exposed to the same painful stimulus. One group experiences a painful stimulus of higher intensity compared to that of the other group. The painful stimuli are physically identical for every subject within the same group and within the standard of previous pain research.
  Participants are then asked to evaluate the painful stimulus they just received according to a self-reported scale (NRS, VAS, gLMS, NRS-MB). Participants are also asked to decide multiple times whether they prefer a larger amount of money and experience the same or more painful stimulus they received before or a smaller amount of money and no (or a less) painful stimulus. The smaller amount of money is progressively increased across choices until it matches the larger amount, similar to multiple price-list methods (MPL) which are standard in economics.
  Arms: Study 1 High-Intensity Group; Study 1 Low-Intensity Group; Study 2 High-Intensity Group; Study 2 Low-Intensity Group; Study 3 Painkiller group; Study 3 Placebo group

SUMMARY:
Pain is a public health challenge around the world. However, there is no single standardized measure of pain, to the point that the estimated prevalence of chronic pain in adults ranges between 2% and 64% depending on the methods and definitions used. Existing measures of pain are known to present several problems and results can be hardly compared between people.

The investigators propose and empirically validate a new, simple method to measure experienced pain in clinical trials. The method provides an objective, cardinal measurement of experienced pain which is comparable between people and the investigators test whether it is better able to measure experienced pain than existing procedures. The investigators test the new method in healthy participants using standard protocols (electrical and heat stimuli). The investigators also aim to validate the measure using a causal manipulation which relies on the administration of a topical analgesic product compared to a placebo.

DETAILED DESCRIPTION:
The aim of this study is to establish and validate the proposed method of measuring pain using different pain stimuli. The investigators correlate these measurements with physiological data such as skin-conductance, heart-rate variability, pupil dilation, and with established measures of pain such as Numeric rating scale (NRS), Visual analog scale (VAS), general Labeled Magnitude Scale (gLMS). In addition, the investigators study the test-retest reliability of our measure of pain and its ability to capture a reduction in experienced pain due to a topical analgesic product compared to a placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years.
* ability and willingness to participate in the study
* declaration of consent
* good English language skills (to ensure understanding of all instructions and the declaration of consent).

Exclusion Criteria:

* inability to give the declaration of consent (e.g. due to linguistic difficulties understanding the study information)
* any neurological disorders
* reduced general health / chronic diseases (e.g. autoimmune disease, severe cardiovascular diseases, insulin-dependent diabetes, severe depression); chronic pain disorders
* pregnancy
* in the week before the experimental session self-reported intake of drugs which could influence pain perception (e.g. cannabis and ADHD medications).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Choices between monetary amounts and painful stimuli | baseline
  Participants' choices between monetary amounts and painful stimuli
self-reported pain ratings according to Numerical Rating Scale (NRS) | baseline
  self-reported pain ratings according to Numerical Rating Scale
self-reported pain ratings according to Visual Analogue Scale (VAS) | baseline
  self-reported pain ratings according to Visual Analogue Scale
self-reported pain ratings according to general Labeled Magnitude Scale (gLMS) | baseline
  self-reported pain ratings according to general Labeled Magnitude Scale
response times | baseline
  Response times relative to participants' choices between monetary amounts and painful stimuli

SECONDARY OUTCOMES:
heart rate variability | baseline
  variation in heat-beat rate in reaction to the painful stimuli.
skin conductance | baseline
  variation in skin conductance in reaction to the painful stimuli.
pupil dilation | baseline
  variation in pupil dilation in reaction to the painful stimuli.

CONTACTS AND LOCATIONS:
Locations (1):
- SNS Laboratory, Zurich, CH, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided